CLINICAL TRIAL: NCT06021054
Title: A Randomized, Double-masked, Placebo-controlled Safety, Tolerability, and Efficacy Study of Veligrotug (VRDN-001), a Humanized Monoclonal Antibody Directed Against the IGF-1 Receptor, in Participants With Chronic Thyroid Eye Disease (TED)
Brief Title: An Efficacy, Safety, and Tolerability Study of Veligrotug (VRDN-001), in Participants With Chronic Thyroid Eye Disease (TED) (THRIVE-2)
Acronym: THRIVE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Viridian Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VRDN-001-301
Record Dates: First submitted 2023-08-25; First posted 2023-09-01 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Thyroid Eye Disease
Keywords: Thyroid Eye Disease; Thyroid-Associated Ophthalmopathy; Dysthyroid Ophthalmopathy; Graves Eye Disease; Graves Orbitopathy; Myopathic Ophthalmopathy; Congestive Ophthalmopathy; Edematous Ophthalmopathy; Infiltrative Ophthalmopathy; TED; Thyroid-Associated Orbitopathy; Graves Disease
MeSH Terms: conditions — Graves Ophthalmopathy; Graves Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Veligrotug (VRDN-001)10 mg/kg (Experimental): Drug: 5 IV Infusions of veligrotug (VRDN-001)10 mg/kg
  Interventions: Drug: Veligrotug (VRDN-001)
- Placebo Drug (Experimental): Placebo Drug: 5 IV Infusions of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Veligrotug (VRDN-001) — Veligrotug (VRDN-001) is a humanized monoclonal antibody directed against the IGF-1 receptor
  Arms: Veligrotug (VRDN-001)10 mg/kg
Drug: Placebo — 5 IV infusions of placebo
  Arms: Placebo Drug

SUMMARY:
This is a clinical trial assessing the efficacy, safety, and tolerability of an investigational drug, veligrotug (VRDN-001), in participants with chronic thyroid eye disease (TED).

DETAILED DESCRIPTION:
This is a randomized (meaning participants will be assigned to study arms by chance), double-masked (meaning study doctor and participant will not know which study arm participant is assigned to), placebo-controlled study that will include participants with chronic TED. The key objectives of this study are to determine if veligrotug (VRDN-001) is efficacious, safe, and tolerable when administered as 5 IV infusions given every 3 weeks for a total of 12 weeks in participants with chronic TED

ELIGIBILITY:
Key Inclusion Criteria:

* Must have moderate to severe chronic TED with documented evidence of ocular symptoms or signs that began greater than 15 months prior to screening
* Must have had a clinical diagnosis of TED, with any CAS (0-7)
* Must agree to use highly effective contraception as specified in the protocol
* Female TED participants must have a negative serum pregnancy test at screening

Key Exclusion Criteria:

* Must not have received prior treatment with another anti-IGF-1R therapy
* Must not have received systemic corticosteroids for any condition, including TED, or selenium within 2 weeks prior to first dose
* Must not have received other immunosuppressive drugs or another investigational agent for any condition, including TED, or any other therapy for TED, within 8 weeks prior to first dose
* Must not have received radioactive iodine (RAI) treatment within 8 weeks prior to first dose
* Must not have a pre-existing ophthalmic condition in the study eye that in the opinion of the study doctor would confound interpretation of the study results
* Must not have had previous orbital irradiation or decompression surgery for TED to the study eye's orbit
* Must not have inflammatory bowel disease
* Have abnormal baseline audiometry Pure Tone Average (PTA) assessment or history of significant (as determined by the Investigator) ear pathology, relevant ear surgery or hearing loss.
* Female TED participants must not be pregnant or lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Proptosis Responder Rate in the most proptotic eye | Week 15
  Proptosis Responder Rate in the most proptotic eye (i.e., reduction of proptosis of ≥2 mm from baseline [without a corresponding increase of ≥2 mm in the other eye]) as measured by exophthalmometer.

SECONDARY OUTCOMES:
Change from baseline in proptosis in the most proptotic eye | Week 15
  Change from baseline in proptosis in the most proptotic eye as measured by exophthalmometer
Proptosis Responder Rate in the most proptotic eye | Week 15
  Change from baseline in proptosis in the most proptotic eye
Clinical Activity Responder Rate in the most proptotic eye | Week 15
  Clinical Activity Responder Rate in the most proptotic eye (i.e., no worsening in CAS from baseline [without a corresponding increase of ≥2 points in the other eye]) as measured by exophthalmometer
Overall Responder Rate in the most proptotic eye | Week 15
  Overall Responder Rate comprised of Proptosis Responder Rate in the most proptotic eye as measured by exophthalmometer and Clinical Activity Responder rate in the most proptotic eye as measured by exophthalmometer
Diplopia Responder Rate | Week 15
  Diplopia Responder Rate (i.e., reduction in Gorman Subjective Diplopia Score of ≥1 from baseline for participants with baseline Gorman Subjective Diplopia Score >0)
Diplopia Resolution Rate | Week 15
  Diplopia Resolution Rate (i.e., reduction in Gorman Subjective Diplopia Score to 0 from baseline for participants with baseline Gorman Subjective Diplopia Score > 0)

CONTACTS AND LOCATIONS:
Locations (57):
- United States (23):
  - Advancing Research International, LLC, Los Angeles, California
  - USC Roski Eye Institute, Los Angeles, California
  - Amy Patel Jain, MD, Newport Beach, California
  - Stanford Byers Eye Institute, Palo Alto, California
  - Cockerham Eye Consultants, PC, San Diego, California
  - Bascom Palmer Eye Institute - Ophthalmology - Miami, Miami, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Northwestern University, Chicago, Illinois
  - Family Eye Physicians, Ltd, Oak Lawn, Illinois
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Michigan State University, Department of Neurology, East Lansing, Michigan
  - Kahana Oculoplastic and Orbital Surgery, Livonia, Michigan
  - Washington University School of Medicine in St Louis - Ophthalmology, St Louis, Missouri
  - Steven Leibowitz, MD., Las Vegas, Nevada
  - Rutgers - New Jersey Medical School, Newark, New Jersey
  - The Center for Eye and Facial Plastic Surgery, Somerset, New Jersey
  - Department of Ophthalmology, University of Pennsylvania, Philadelphia, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Baylor College of Medicine (BCM) - Ophthalmology, Houston, Texas
  - Neuro Eye Clinical Trials, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Harborview Medical Center, Seattle, Washington
- North Shore Private Hospital, Saint Leonards, New South Wales, Australia
- France (4):
  - CHU Angers, Angers
  - CHU de Bordeaux - Hôpital Saint-André, Bordeaux
  - Centre Hospitalier Universitaire De Nantes - G. R. Laennec, Nantes
  - CH Nice, Nice
- Germany (4):
  - Charité - Universitätsmedizin Berlin KöR, Berlin
  - Universitätsklinikum Essen AöR, Essen
  - University Medical Center Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Göttingen
- Hungary (3):
  - Budapest Retina Intezet, Budapest
  - Ganglion Orvosi Kozpont, Pécs
  - Pecsi Tudomanyegyetem Klinikai Kozpont Szemeszeti Klinika, Pécs
- Poland (5):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Oculomedica Sp. z o.o., Bialystok
  - Optimum Profesorskie Centrum Okulistyki Sp. z o.o., Gdansk
  - Centrum Medyczne Pulawska Sp. z o.o., Piaseczno
  - Centrum Medyczne Piasta 47 sp. z o.o., Wałbrzych
- Spain (8):
  - Complexo Hospitalario Universitario de Santiago-Hospital Médico-Cirúrxico de Conxo, A Coruña
  - Centro de Oftalmologia Barraquer (Barraquer Ophthalmology Centre), Barcelona
  - Hospital La Arruzafa, Córdoba
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen De La Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Y Politécnico La Fe, Valencia
  - Hospital Unviersitario Miguel Servet, Zaragoza
- Turkey (Türkiye) (4):
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Gazi University Medical Faculty Hospital, Ankara
  - Akdeniz University Medical Faculty Hospital, Antalya
  - Marmara University Faculty of Medicine, Istanbul
- United Kingdom (5):
  - Moorfield's Eye Hospital, London
  - Imperial College Healthcare NHS Trust - Western eye Hospital, London
  - Guy's and St. Thomas NHS Trust, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - University Hospital Southampton NHS Foundation Trust, Southampton